CLINICAL TRIAL: NCT01542151
Title: Effects of Sleep, Fatigue, and Timing of Post-dates Inductions Among Nulliparas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: TimeIOL
Record Dates: First submitted 2012-01-24; First posted 2012-03-02 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Pregnancy, Prolonged
Keywords: Labor, induced; Sleep; Fatigue; Patient satisfaction; Circadian rhythm
MeSH Terms: conditions — Pregnancy, Prolonged; Fatigue; Patient Satisfaction | interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morning (Active Comparator): Women randomized to a labor induction in the morning between 0600 and 1000.
  Interventions: Other: Time of labor induction
- Evening (Experimental): Women randomized to a labor induction begun in the evening between 1700-2100
  Interventions: Other: Time of labor induction

INTERVENTIONS:
Other: Time of labor induction — Assigned time of labor induction - morning or evening
  Other Names: Labor, induced

SUMMARY:
This randomized clinical trial will examine if there are any differences between post-dates inductions (inductions after 40 weeks of pregnancy) begun in the morning compared to the evening for first-time mothers. Sleep and fatigue measures will be measured to see if they differ by time of induction. Other measures will include the rate of births within 24 hours of admission, length of labor, use of labor analgesics, and method of delivery.

DETAILED DESCRIPTION:
Randomized clinical trial of first-time pregnant women requiring post-dates induction (induction after 40 weeks gestation). Women will be randomized to a labor induction time in the morning or the evening. On hospital admission once women have signed the study consent, they will complete sleep questionnaires and a fatigue assessment. Fatigue and sleep time assessments will subsequently done by the study subject every 4 hours until women enter active labor. At the onset of active labor, assessments will stop. Labor outcomes and patient satisfaction will be obtained once women deliver.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at 40 weeks gestation or more
* Nulliparous
* 14 years old or older
* English or Spanish speaking
* Healthy maternal status
* Labor induction able to be scheduled

Exclusion Criteria:

* Less than 40 weeks gestation
* Multiparous
* Younger than 14 years old
* Not able to speak or write in English or Spanish
* Fetal or maternal status requires immediate induction

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Birth within 24 hours of induction | Day 1
  Calculate proportion of women delivering within 24 hours of the start of labor induction between the two groups

SECONDARY OUTCOMES:
Cesarean rate | Day 1
  Compare cesarean rates between the two groups
Change in fatigue scores | Day 1
  Differences in Fatigue Visual Analog Scales from admission to active labor between the two groups.
Change in hand grip strength | Day 1
  Differences in change in hand grip strength from admission to active labor between the two groups.
St. Mary's Sleep scale | Prebaseline: Baseline - 12-24 hours
  Differences in St. Mary's Sleep scores on admission between the two groups.
Labor and birth satisfaction | Day 2
  Differences in Labor and Birth Satisfaction between the two groups.
Morning-evening chronotype | Day 1
  Correlation between Horne-Osteberg Morning-Eveningness chronotype and birth within 24 hours of start of induction.
Sleep Quality | Prebaseline: Baseline - 30 days
  Correlation between sleep quality in the one month prior to admission measured with the Pittsburgh Sleep Quality Index and birth within 24 hours of start of induction.
Length of time to labor intervention | Day 1
  Measure differences between groups between length of time from admission to different labor interventions e.g., rupture of membranes, analgesia - IV or epidural
Neonatal outcomes | Day 1
  Differences between groups on neonatal outcomes such as 5 minute Apgar scores and admission to neonatal intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Barger, PhD, Principal Investigator — University of Clifornia, San Francisco
Locations (1):
- Community Medicall Center, Fresno, California, United States